CLINICAL TRIAL: NCT00197613
Title: The Adult Antiretroviral Treatment and Resistance Study (Tshepo)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Princess Marina Hospital, Botswana (Unknown); Botswana Ministry of Health (Other Government); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Richard Marlink, Professor of the Practice of Public Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: HSC #0110THEA
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: AIDS; HIV Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Zidovudine; Lamivudine; Nevirapine; efavirenz; Didanosine; Fumigant 93; Stavudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: (A) zidovudine, lamivudine and nevirapine
Drug: (B) zidovudine, lamivudine and efavirenz
Drug: (C) zidovudine, didanosine, and nevirapine
Drug: (D) zidovudine, didanosine, and efavirenz
Drug: (E) stavudine, lamivudine, and nevirapine
Drug: (F) stavudine, lamivudine and efavirenz
Procedure: Adherence Strategy Standard of Care (SOC)
Procedure: Adherence Strategy Community-Based DOT

SUMMARY:
The "Adult Antiretroviral Treatment and Resistance Study," hereafter referred to as "The Tshepo Study," is the first large-scale research study of antiretroviral therapy to treat AIDS and HIV infection in Botswana. The Tshepo Study is an open-label, randomized study comparing: (1) the rate of development and specific types of drug resistance mutations with various antiretroviral combination therapies to HIV-1C, the subtype of HIV found in southern Africa, and (2) the short and long-term effectiveness of two operational modifications of Directly Observed Therapy (DOT) medication adherence strategies for antiretroviral therapy. Specifically, treatment follow-up via the Standard of Care, the national standard of care as it evolves in Botswana, with intensive clinic-based follow up including regular adherence education sessions, will be compared to Community-Based Directly Observed Therapy (Com-DOT). Com-DOT involves the SOC with added community or family-based DOT. This Com-DOT component would involve a trained, community or family-based Medication Partner ("mopati") who observes the patient take his or medications daily.

ELIGIBILITY:
Inclusion Criteria:(1) HIV infection indicated by (a) positive ELISA in two separate blood samples, the second no more than eight weeks prior to randomization), (b) CD4 cell count of less than 200 cells/ml OR CD4 cell count between 201-350 with plasma HIV-1 RNA level of greater than 55,000 copies/ml, (c) Karnofsky (performance) score greater than or equal to 50; (2) no history of previous antiretroviral therapy, except for zidovudine and/or single-dose nevirapine administered during pregnancy to prevent mother-to-child HIV transmission of HIV-1; (3) baseline hemoglobin of greater than or equal to 8.0 g/dl (4) baseline absolute neutrophil count greater than or equal to 1000 cells/mm3 (5) baseline serum creatinine level less than 200 micromol/L (6) baseline SGPT(ALT) less than 205 U/L and SGOT (AST) less than 170 U/L (7) baseline alkaline phosphatase level less than or equal to 330 U/L etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2002-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to Virological failure, time to grade 3 or higher toxicity.

SECONDARY OUTCOMES:
Time to drug resistance, rates of point mutations at virological failure, adherence to study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marlink, MD, Principal Investigator — Harvard School of Public Health AIDS Initiative
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana